CLINICAL TRIAL: NCT01402037
Title: Relation Between Residual Beta Cell Function and Glycemic Variability in (Pre) Type 1 Diabetes.
Brief Title: Beta Cell Function in (Pre)Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ-VUB (Other)
Collaborators: Vrije Universiteit Brussel (Other); University Hospital, Ghent (Other); University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Bart Keymeulen, MD PhD, AZ-VUB
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KD_BF_02
Record Dates: First submitted 2011-07-07; First posted 2011-07-26 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; Prevention; First degree relatives; High risk for type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucose; Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- NDP 12-39 y (Other): In newly diagnosed patients a hyperglycemic clamp tests will be performed within 4 weeks after diagnosis and 6, 12, 18 and 24 months later in 40 patients. The clamp will not be carried out in participants who became Cpeptide negative (defined as AUC C-peptide ≤ 0.03 nmol/L x min.) at a previous visit. HbA1c will be determined at the day of the clamp and glycemic variability during 5 days starting immediately after the clamp procedure. Insulin requirements and severe hypoglycemia (defined as an episode in which a patient required the assistance of another person and which was associated with a blood level of < 50 mg/dL or prompt recovery following intravenous glucose, glucagon or oral carbohydrate) will be recorded
  Interventions: Drug: Glucose; Device: Continuous glucose monitoring
- NDP 5-12 y (Other): Ten childhood-onset patients (under age 12) will be tested for 5 days with CGM (without clamp) and their glycemic variability compared with that of 10 patients aged 12-17 years at diagnosis.
  Interventions: Device: Continuous glucose monitoring
- FDR 12-39 y (Other): In first degree relatives of type 1 diabetes patients a hyperglycemic clamp tests will be performed at inclusion and 6, 12, 18 and 24 months later in 40 high-risk first-degree relatives (see previous definition) with a non-diabetic OGTT performed 1 to 2 weeks before the clamp procedure. An OGTT result suggestive of diabetes will be confirmed and the relative will be offered participation in the patient arm of the study. HbA1c will be determined at the day of the OGTT and glycemic variability during the 5 days preceding the OGTT procedure.
  Interventions: Drug: Glucose; Device: Continuous glucose monitoring
- FDR 5-12 y (Other): Ten high-risk first-degree relatives (see criteria) aged 5 to 12 years will also be tested for CGM and their results correlated with beta-cell function derived from a "mini-clamp" procedure (first 10 min. C-peptide release in hyperglycemic clamp) and results (CGM and first clamp phase) from relatives aged 12-17 years.
  Interventions: Drug: Glucose; Device: Continuous glucose monitoring

INTERVENTIONS:
Drug: Glucose — Glucose 20% intravenous
  Other Names: Stimulated glucose
  Arms: FDR 12-39 y; FDR 5-12 y; NDP 12-39 y
Device: Continuous glucose monitoring — Blood glucose profiles: during 5 days glucose profiles will be determined by seven-point self-monitoring of blood glucose (SMBG) (pre-breakfast: assumed time 7 am, post-breakfast: 8.30 am, pre-lunch: 12 am, post-lunch: 1.30 pm, pre-supper: 6 am, post-supper: 7.30 pm, bedtime: 10 pm) and by continuous glucose monitoring (CGM). Participants will be blinded for the CGM results.
  Other Names: CGM

SUMMARY:
Increased glycemic variability has been proposed as an independent predictor of hypoglycemia in diabetic patients. Likewise, episodes of dysglycemia have been found to be predictive of diabetes in antibodypositive nondiabetic individuals. We hypothesise that an in-depth observational study comparing state-of-the-art measures of functional beta cell mass and glycemic variability will specify the relationship between both variables over a broad range of residual function and will identify treatment goals for functional beta cell mass to be reached in future beta cell therapy trials in order to avoid frequent hypoglycemia in patients and dysglycemia in risk groups. The available expertise and infrastructure (see background and (inter)national context) place the promoters of the present project in a unique position to carry out the planned experiments and support their feasibility.

DETAILED DESCRIPTION:
The established clinical network and the developed dynamic function tests and biological markers provide us with the unique opportunity to identify sufficiently large groups of high-risk first-degree relatives (> 50% risk of diabetes) of a proband with type 1 diabetes and of recent-onset type 1 diabetic patients with the overall aim to investigate the correlation between functional beta cell mass and glycemic variability in relation to metabolic outcome in order to determine thresholds of residual function below which:

1. glucose tolerance starts to decline sharply in relatives
2. the risk of deteriorating metabolic control and (severe) hypoglycemic events strongly increases in patients

To this effect we will:

1. measure and follow over a two-year period

   1. the functional beta cell mass of participants as determined by AUC C-peptide release - the preferred outcome measure in type 1 diabetes trials during hyperglycemic clamp test
   2. the participants' within- and between-day glycemic variability as determined by seven point selfmonitoring of blood glucose (SMBG) and continuous glucose monitoring (CGM) during 5 days preceding each clamp procedure
2. perform oral glucose tolerance tests (OGTTs; only in relatives), determine HbA1c levels centrally (relatives and patients) and record insulin requirements and hypoglycemic episodes (in patients) Our previous experiments have documented that the selected patients and relatives (see workplan) display large inter-individual differences in functional beta cell mass (ranging anywhere between control values and < 10% of controls) allowing to study glycemic variability as a function of residual cell function over a large range of values. They also illustrate that the recruitment capacity of the clinical network and the acceptance rate and compliance of the patients and relatives for the clamp procedure is high and sufficient to carry out the planned experiments.

ELIGIBILITY:
Inclusion Criteria:

Type 1 diabetic patients:

1. aged 12-39 years at diagnosis
2. treated with insulin for less than 4 weeks
3. optimally treated with intensified insulin treatment: minimal three preprandial injections of ultra-rapidly acting analogs and one evening injection of long-acting insulin (Lantus®, Sanofi Aventis)
4. positive for autoantibodies against insulin (IAA-sampled within the first week of insulin treatment), 65kDa glutamate decarboxylase (GADA), IA-2 protein (IA-2A) and/or zinc transporter 8 (ZnT8A)

First-degree relatives:

1. aged 12-39 years at inclusion
2. sibling or offspring of a type 1 diabetic patient diagnosed before age 35 or between age 35 and 50 with in addition a body mass index < 28 kg/m2 and an initial insulin dose > 0.25 U.kg -1.d-1
3. > 50% risk of diabetes within 5 years as indicated by positivity for at least 2 diabetes antibodies including IA-2A and/or ZnT8A in absence of protective HLA-DQ genotypes (6)

Exclusion Criteria:

* pregnancy or lactation in women
* use of illicit drugs or overconsumption of alcohol or history of drug or alcohol abuse
* being legally incapacitated, having significant emotional problems at the time of the study, or having a history of psychiatric disorders
* having received antidepressant medications during the last 6 months
* treatment with immune modulating or diabetogenic medication (such as corticosteroids)
* history of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risks to the subjects
* patients not treated with Lantus as insulin therapy.

Ages: 5 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
evaluate the hyperglycemic clamp to measure the functional beta cell mass test | 2 years
  to measure the functional beta cell mass of participants as determined by AUC C-peptide release during hyperglycemic clamp test

SECONDARY OUTCOMES:
Follow up of OGTT's and HbA1c levels in high risk first degree relatives and patients | 2 years
  2) perform oral glucose tolerance tests (OGTTs; only in relatives), determine HbA1c levels centrally (relatives and patients) and record insulin requirements and hypoglycemic episodes (in patients)
evaluate the continuous glucose monitoring to measure within- and between-day glycemic variability | 2 years
  to measure within- and between-day glycemic variability as determined by seven point selfmonitoring of blood glucose (SMBG) and continuous glucose monitoring (CGM) during 5 days preceding each clamp procedure

CONTACTS AND LOCATIONS:
Overall Officials: Frans K Gorus, MD. PhD., Principal Investigator — UZ Brussels
Locations (3):
- Belgium (3):
  - UZ Brussels, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent